CLINICAL TRIAL: NCT02590614
Title: Genetic, Dietary and Environmental Influences on Vitamin D Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Robin Taylor Wilson, Associate Professor of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 209517-REV1
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 800 IU Vitamin D (Experimental): Participants will be taking 800 IU/d of vitamin D3 for two months
  Interventions: Dietary Supplement: 800 IU Vitamin D
- Placebo (Placebo Comparator): Placebo made by Vital Nutrients, Inc. to look exactly like the 800 IU/d caplets by the same company.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 800 IU Vitamin D — Among the cross-sectional study participants, a subset is randomly selected and matched based on genetic ancestry, and randomized to the intervention group.
  Other Names: Vital Nutrients
  Arms: 800 IU Vitamin D
Dietary Supplement: Placebo — Among the cross-sectional study participants, a subset is randomly selected and matched based on genetic ancestry, and randomized to the placebo group
  Other Names: Vital Nutrients Placebo
  Arms: Placebo

SUMMARY:
Determine differences in serum vitamin D metabolism by genetic ancestry.

DETAILED DESCRIPTION:
Vitamin D metabolites are well-recognized to stop cancer cell growth in culture. However, a clear definition of a sufficient level of serum vitamin D (currently measured as 25(OH)D) for disease prevention has been hampered by inconsistent results from both observational studies and randomized clinical trials. Observational cancer studies report both increased and reduced risks of cancer in subjects with higher serum levels of 25(OH)D, while large randomized trials report no significant benefit of vitamin D supplementation for breast cancer (incidence), colon cancer (incidence and mortality), lung cancer (mortality), or benign proliferative breast disease.

The 25(OH)D metabolite of vitamin D (comprised of 25(OH)D3 and 25(OH)D2), is the principal hydroxylated metabolite in serum and is considered a reasonable functional biomarker of vitamin D status. This is because, although subject to seasonal variation, multiple measurements in the same individual are relatively consistent over time. The most biologically active vitamin D metabolite is 1,25(OH)2D3, and may therefore be the most relevant to long-term health outcomes. Nonetheless, 1,25(OH)2D3 is not frequently used as a biomarker in epidemiologic studies as it displays diurnal variation and has a short in vivo half life.

Notably, in vivo treatment with 1,25(OH)2D3 is associated with increased metabolic clearance of 25(OH)D3, decreased serum 25(OH)D3 levels, and a higher 25(OH)D3 to 24,25(OH)2D3 conversion rate in humans and animals. This suggests that use of 25(OH)D as single biomarker of vitamin D status does not fully capture the entire picture. Paradoxically, one individual may be classified with 'low' 25(OH)D as a consequence of low dietary intake and little sun exposure while yet another individual classified with 'low' 25(OH)D may actually have a higher concentration of the 1,25(OH)2D3 metabolite-possibly due to genetic differences in enzymes that metabolize vitamin D (CYP2R1, CYP27B1, and CYP24A1).

Genome-wide and candidate gene association studies of serum 25(OH)D levels have suggested a role of single nucleotide polymorphisms (SNPs) near the vitamin D binding protein (GC) and CYP2R1. However, the investigators and others have shown that serum 25(OH)D levels are also associated with genetic ancestry. Because existing studies do not adjust for genetic ancestry and the function of these SNPs have yet to be established, it is not known whether these SNPs actually play a role or whether these may be spurious associations due to ancestral background (i.e., population stratification), correlations with truly causal SNPs, or to random chance. In addition, because of the number of SNPs that must be distinguished, genome-wide studies do not capture regions with high homology or sequence repeats, such as the promoter region of CYP24A1 which has a higher guanine-cytosine content. Improved classification of 'low' 25(OH)D levels within the context of a particular genetic background through identification of "rapid" versus "slow" vitamin D metabolizers will likely have important implications for cancer risk.

It is well-recognized that individuals with African Ancestry have substantially lower (~2-fold) serum 25(OH)D levels compared with other racial/ethnic groups. These differences have been attributed primarily to skin pigmentation. However, the relation between serum 25(OH)D levels and health outcomes is complex and involves a number of variables including diet, sun exposure and hormone status. For example, despite lower average dietary intake of both calcium and vitamin D, and lower serum 25(OH)D levels, African Americans have higher bone mineral density and a 3-fold lower risk of hip fracture relative to European Americans. There are some lines of evidence which suggest that African Americans may have comparatively higher circulating levels of 1,25(OH)2D3, although most studies are small and do not account for age and/or diurnal variation, and this may explain why other studies report no difference.

Among Europeans alone, a moderately high heritability of serum 25(OH)D levels (~50 to 70% for 25(OH)D) has been observed, as well as associations between 25(OH)D and several genetic polymorphisms in vitamin D metabolizing enzymes, although the functional consequences of these polymorphisms are not known. Small and large clinical trials among healthy individuals have also noted substantial inter-individual differences(as much as 5-fold) in the increases of serum 25(OH)D levels among participants given the same oral dose of vitamin D, the same minimal erythema dose (MED) of UV-B light, or the same dose of UV light. The importance of understanding inter-individual differences in vitamin D synthesis, metabolism and effect have been underscored by results from high dose randomized trials reporting that those in the vitamin D supplementation groups experienced a 31% higher bone fracture incidence, and significantly lower prostate cancer survival. There is a clear need to understand individual differences in the metabolism of vitamin D before future high dose trials proceed.

Previous Data: Studies by the investigators' lab and others have identified significant racial/ethnic differences in the frequency of variants in genes responsible for vitamin D metabolism (i.e., CYP2R1, CYP27B1 and CYP24A1). In collaboration with the Pike Laboratory (University of Wisconsin), the investigators' laboratory has identified several novel genetic variants in recently identified regulatory regions of the gene which encodes for the major vitamin D catabolic enzyme (CYP24A1).

Study Rationale:The role/function of these polymorphisms has not been tested in either epidemiologic association studies or in cell-based assays. It will be important to complement genetic association studies with multiple types of molecular assays that can tell a consistent story about the likely role of a particular genetic variant.

The investigators hypothesize that there is a significant influence of genetic variants on serum vitamin D metabolism that is independent of genetic ancestry, skin melanin content, sunlight exposure and dietary/supplement intake.

Study Objectives:A small randomized study in healthy subjects will investigate temporal changes in the balance of metabolites (25(OH)D3, 25(OH)D2, 24,25(OH)2D3 and 1,25(OH)2D3) following a two-month course of vitamin D3 (800 IU/d).

This study overcomes limitations of existing genetic association studies that may report spurious results due to lack of control for genetic ancestry, skin reflectance, collection of blood specimens during summer months, or the use of assays that do not distinguish 25(OH)D2 and 25(OH)D3. The advantages of this study are: 1) a matched design that incorporates temporal assessment of vitamin D metabolism, 2) genetic Ancestry Informative Markers (AIMs), 3) melanin skin index, 4) a sensitive and reliable assay for four serum vitamin D metabolites, and 5) functional molecular assays related to specific genetic polymorphisms.

The investigators' research addresses one of the major research gaps in the understanding of the health-related benefits of vitamin D identified by a recent Institute of Medicine Review. While vitamin D metabolites have significant anti-cancer properties, a better understanding of the genetic influences upon vitamin D metabolism is needed in order to improve the identification of cancer risks associated with vitamin D.

Study Design: This study employs two designs-first a cross-sectional study of participants is selected.

Among the cross-sectional study participants, a subset is randomly selected and matched based on genetic ancestry, and randomized to either the intervention (800 IU/day of vitamin d) or placebo group.

Statistical Plan:In the first portion of this study, an estimated 400 participants will be screened to determine eligibility. Eligibility screening will be completed online through RedCap.

In the second portion of this study, participants randomly chosen from the original 400 for the Supplement Intervention Study will be asked to complete 3 additional blood draws at Week 0, 4 and 8 of the Supplement Intervention Study (N=64).

The 64 Supplement Intervention study participants will be randomly chosen from the eligible participants in the first part of the study (n=400). Sample size calculations were performed by Dr. Vernon Chinchilli in order to estimate the number of participants that the investigators would need in order to detect differences in their vitamin D levels. The investigators accounted for loss-to-follow-up and normal withdrawal from the study.

NOTE:

The total participants that will get screened has been changed (from the original AICR grant) and revised in the budget from 300 to 400 participants. The investigators made this revision because the investigators decided that loss to follow-up may be higher than the originally estimated 10%. The investigators then estimated that loss to follow-up may actually be closer to 20%. This proportional difference was calculated from the investigators' original estimate of 52 to 64 (which is about 24% increase in participants) and was revised also to increase the amount of participants that the investigators will screen from the original 300 to an estimated 372 (determined proportionally with a 24% increase). The investigators went ahead and assumed that the upper limit may include 400 participants so that the investigators can end up with 64 participants in the supplementation trial.

The investigators will conduct an intention-to-treat analysis to analyze differences in the serum level of vitamin D metabolites and vitamin D metabolite ratios within supplement and placebo group pairs at times 0, 1 month and 2 months. Differences in the pairwise log concentration of metabolites and log metabolite ratios will be tested by Wilcoxon Signed-Rank Tests and linear mixed-effect models (SAS Proc Mixed) using restricted maximum likelihood estimation to account for one time point as well as repeated measures of vitamin D metabolites. Potential confounding and effect modification by dietary intake of vitamin D will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy African American and Caucasian adult volunteers
2. Aged 18 to 35
3. At least 50% African American or at least 50% Caucasian
4. Willing to take a vitamin D supplement for two months
5. Willing to attend monthly visits to the clinic for blood draw and vital check
6. Willing to refrain from taking other dietary supplements including herbal supplements, multi-vitamins and vitamin D supplements other than the supplements provided in the trial.
7. Willing to avoid tanning bed use during the above mentioned period.
8. Willing to avoid extensive use of analgesics and have the consumption of the following drugs recorded: Acetaminophen, Celecoxib, Codeine, Fentanyl, any antibiotics, and Hormonal IUD.

Exclusion Criteria:

1. Participants with a fever (100 degrees F or higher) at the time of the visit
2. Participants with severe chronic disease (i.e., chronic kidney disease, cirrhosis of the liver, heart attack, HIV/AIDS, alcoholism, hemophilia, sickle cell disease, or other serious underlying illness that prevents blood donation),
3. Participants that have received radiation therapy or chemotherapy within the past 4 weeks,
4. Participants with any of the following on the upper right arm: rashes, a cast, swelling, paralysis, open sores or wounds.
5. Individuals with blindness and/or deafness
6. Pregnant participants will be excluded from the study.
7. Participants taking any of the following medications will be excluded from the study:

   1. Long-term antibiotic use: Clarithromycin, Ciprofloxacin, Erythromycin, Telithromycin, Nafcillin
   2. Chemotherapy for cancer
   3. Prescription vitamin supplement
   4. Anti-convulsants: Carbamazepine, Pentobarbital, Phenobarbital, Phenytoin, Primidone, Fosphenytoin
   5. Erectile dysfunction drugs: sildenafil, vardenafil, tadalafil
   6. Immunosuppressants: Tacrolimus, Cyclosporine A, Sirolimus, Mycophenolate, Glucocorticoids (like Dexamethasone)
   7. Proton-pump inhibitors: omeprazole lansoprazole, dexlansoprazole, rabeprazole, pantoprazole, and esomeprazole
   8. Calcium Channel Blockers: nifedipine, felodipine, isradipine, nicardipine, nifedipine, nisoldipine, amlodipine, lacidipine, Verapamil, diltiazem
   9. Diuretics : furosemide, bumetanide, torsemide, ethacrynic acid, amiloride, triamterene, spironolactone, eplerenone,
   10. Statins: lovastatin, simvastatin, atorvastatin, Pravastatin, fluvastatin, rosuvastatin, pitavastatin, Orlistat (Xenical, Alli),
   11. Anti-fungal: Itraconazole, Ketoconazole, Posaconazole, Voriconazole, Fluconazole, Isavuconazole (isavuconazonium sulfate) Clotrimazole
   12. HIV protease inhibitors and other anti-retrovirals : Atazanavir, Boceprevir, Darunavir, Indinavir, Lopinavir, Nelfinavir, Ombitasvirparitaprevirritonavir, Ombitasvirparitaprevirritonavir plus dasabuvir, Ritonavir and ritonavir containing coformulations, Saquinavir, Telaprevir
   13. TB medications: Rifabutin, Rifampin (rifampicin), Rifapentine
   14. As well as CYP3A4 inhibitors including: Ceritinib, Cobicistat and cobicistat containing coformulations, Idelalisib, Nefazodone, Amiodarone, Aprepitant, Cimetidine, Conivaptan, Crizotinib, Delavirdine, Desipramine, Dronedarone, Fosaprepitant Mifepristone, Netupitant, Nilotinib, and Tibolone
   15. As well as CYP3A4 inducers including: Dexamethasone, Enzalutamide, Lumacaftor, Mitotane, St. John's wort, Bexarotene, Bosentan, Dabrafenib, Efavirenz, Eslicarbazepine, Etravirine, Modafinil
   16. Other drugs that will cause a participant to be excluded include: Cholestyramine, Ferric carboxymaltose (treatment of iron deficiency anemia), Dapsone, Metformin

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 412 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of 25(OH)D3 | Three month change
  Differences in the increase in fasting serum levels of vitamin D metabolite 25(OH)D3 between African American and European American ancestry pairs will be determined at 0, 1 and 2 months.
Serum concentrations of 24,25(OH)2D3 | Three month change
  Differences in the increase in fasting serum levels of vitamin D metabolite 24,25(OH)D3 between African American and European American ancestry pairs will be determined at 0, 1 and 2 months.
Serum concentrations of 1,25(OH)2D3 | Three month change
  Differences in the increase in fasting serum levels of vitamin D metabolite 1,25(OH)D3 between African American and European American ancestry pairs will be determined at 0, 1 and 2 months.
Metabolite Ratio | Three months
  Difference in the upstream to downstream vitamin D metabolite ratios (24,25(OH)2D3 to 25(OH)D3 and 1,25(OH)2D3 to 25(OH)D3) between African American and European American ancestry pairs will be determined at 0, 1 and 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robin T Wilson, PhD, Principal Investigator — Penn State Hershey, Department of Public Health Sciences
Locations (1):
- Penn State Clinical Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Ahn J, Yu K, Stolzenberg-Solomon R, Simon KC, McCullough ML, Gallicchio L, Jacobs EJ, Ascherio A, Helzlsouer K, Jacobs KB, Li Q, Weinstein SJ, Purdue M, Virtamo J, Horst R, Wheeler W, Chanock S, Hunter DJ, Hayes RB, Kraft P, Albanes D. Genome-wide association study of circulating vitamin D levels. Hum Mol Genet. 2010 Jul 1;19(13):2739-45. doi: 10.1093/hmg/ddq155. Epub 2010 Apr 23. PMID 20418485
- [Background] Al-Delaimy WK, Jansen EH, Peeters PH, van der Laan JD, van Noord PA, Boshuizen HC, van der Schouw YT, Jenab M, Ferrari P, Bueno-de-Mesquita HB. Reliability of biomarkers of iron status, blood lipids, oxidative stress, vitamin D, C-reactive protein and fructosamine in two Dutch cohorts. Biomarkers. 2006 Jul-Aug;11(4):370-82. doi: 10.1080/13547500600799748. PMID 16908443
- [Background] Aronov PA, Hall LM, Dettmer K, Stephensen CB, Hammock BD. Metabolic profiling of major vitamin D metabolites using Diels-Alder derivatization and ultra-performance liquid chromatography-tandem mass spectrometry. Anal Bioanal Chem. 2008 Jul;391(5):1917-30. doi: 10.1007/s00216-008-2095-8. Epub 2008 Apr 24. PMID 18437365
- [Background] Barnholtz-Sloan JS, McEvoy B, Shriver MD, Rebbeck TR. Ancestry estimation and correction for population stratification in molecular epidemiologic association studies. Cancer Epidemiol Biomarkers Prev. 2008 Mar;17(3):471-7. doi: 10.1158/1055-9965.EPI-07-0491. No abstract available. PMID 18349264
- [Background] Barnholtz-Sloan JS, Shetty PB, Guan X, Nyante SJ, Luo J, Brennan DJ, Millikan RC. FGFR2 and other loci identified in genome-wide association studies are associated with breast cancer in African-American and younger women. Carcinogenesis. 2010 Aug;31(8):1417-23. doi: 10.1093/carcin/bgq128. Epub 2010 Jun 16. PMID 20554749
- [Background] Bell NH, Shaw S, Turner RT. Evidence that 1,25-dihydroxyvitamin D3 inhibits the hepatic production of 25-hydroxyvitamin D in man. J Clin Invest. 1984 Oct;74(4):1540-4. doi: 10.1172/JCI111568. PMID 6332830
- [Background] Birlea SA, Costin GE, Norris DA. Cellular and molecular mechanisms involved in the action of vitamin D analogs targeting vitiligo depigmentation. Curr Drug Targets. 2008 Apr;9(4):345-59. doi: 10.2174/138945008783954970. PMID 18393827
- [Background] Boyan BD, Hurst-Kennedy J, Denison TA, Schwartz Z. 24R,25-dihydroxyvitamin D3 [24R,25(OH)2D3] controls growth plate development by inhibiting apoptosis in the reserve zone and stimulating response to 1alpha,25(OH)2D3 in hypertrophic cells. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):212-6. doi: 10.1016/j.jsbmb.2010.03.057. Epub 2010 Mar 20. PMID 20307662
- [Background] Braun MM, Helzlsouer KJ, Hollis BW, Comstock GW. Colon cancer and serum vitamin D metabolite levels 10-17 years prior to diagnosis. Am J Epidemiol. 1995 Sep 15;142(6):608-11. doi: 10.1093/oxfordjournals.aje.a117682. PMID 7653469
- [Background] Brazerol WF, McPhee AJ, Mimouni F, Specker BL, Tsang RC. Serial ultraviolet B exposure and serum 25 hydroxyvitamin D response in young adult American blacks and whites: no racial differences. J Am Coll Nutr. 1988 Apr;7(2):111-8. doi: 10.1080/07315724.1988.10720227. PMID 3361035
- [Background] Brouwer DA, van Beek J, Ferwerda H, Brugman AM, van der Klis FR, van der Heiden HJ, Muskiet FA. Rat adipose tissue rapidly accumulates and slowly releases an orally-administered high vitamin D dose. Br J Nutr. 1998 Jun;79(6):527-32. doi: 10.1079/bjn19980091. PMID 9771340
- [Background] Bu FX, Armas L, Lappe J, Zhou Y, Gao G, Wang HW, Recker R, Zhao LJ. Comprehensive association analysis of nine candidate genes with serum 25-hydroxy vitamin D levels among healthy Caucasian subjects. Hum Genet. 2010 Nov;128(5):549-56. doi: 10.1007/s00439-010-0881-9. Epub 2010 Sep 1. PMID 20809279
- [Background] Chen TC. Photobiology of Vitamin D. In: Holick MF, ed. Vitamin D: Physiology, Molecular Biology, and Clinical Implications. Towtowa, NJ: Humana Press, Inc.; 1999.
- [Background] Chlebowski RT, Johnson KC, Kooperberg C, Pettinger M, Wactawski-Wende J, Rohan T, Rossouw J, Lane D, O'Sullivan MJ, Yasmeen S, Hiatt RA, Shikany JM, Vitolins M, Khandekar J, Hubbell FA; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of breast cancer. J Natl Cancer Inst. 2008 Nov 19;100(22):1581-91. doi: 10.1093/jnci/djn360. Epub 2008 Nov 11. PMID 19001601
- [Background] Chung M, Balk EM, Brendel M, Ip S, Lau J, Lee J, Lichtenstein A, Patel K, Raman G, Tatsioni A, Terasawa T, Trikalinos TA. Vitamin D and calcium: a systematic review of health outcomes. Evid Rep Technol Assess (Full Rep). 2009 Aug;(183):1-420. PMID 20629479
- [Background] Clarys P, Alewaeters K, Lambrecht R, Barel AO. Skin color measurements: comparison between three instruments: the Chromameter(R), the DermaSpectrometer(R) and the Mexameter(R). Skin Res Technol. 2000 Nov;6(4):230-238. doi: 10.1034/j.1600-0846.2000.006004230.x. PMID 11428962
- [Background] De Haes P, Garmyn M, Carmeliet G, Degreef H, Vantieghem K, Bouillon R, Segaert S. Molecular pathways involved in the anti-apoptotic effect of 1,25-dihydroxyvitamin D3 in primary human keratinocytes. J Cell Biochem. 2004 Nov 15;93(5):951-67. doi: 10.1002/jcb.20227. PMID 15389877
- [Background] Feskanich D, Ma J, Fuchs CS, Kirkner GJ, Hankinson SE, Hollis BW, Giovannucci EL. Plasma vitamin D metabolites and risk of colorectal cancer in women. Cancer Epidemiol Biomarkers Prev. 2004 Sep;13(9):1502-8. PMID 15342452
- [Background] Freedman DM, Looker AC, Abnet CC, Linet MS, Graubard BI. Serum 25-hydroxyvitamin D and cancer mortality in the NHANES III study (1988-2006). Cancer Res. 2010 Nov 1;70(21):8587-97. doi: 10.1158/0008-5472.CAN-10-1420. Epub 2010 Sep 16. PMID 20847342
- [Background] Galsky MD, Vogelzang NJ. Docetaxel-based combination therapy for castration-resistant prostate cancer. Ann Oncol. 2010 Nov;21(11):2135-2144. doi: 10.1093/annonc/mdq050. Epub 2010 Mar 29. PMID 20351071
- [Background] Haddad JG, Matsuoka LY, Hollis BW, Hu YZ, Wortsman J. Human plasma transport of vitamin D after its endogenous synthesis. J Clin Invest. 1993 Jun;91(6):2552-5. doi: 10.1172/JCI116492. PMID 8390483
- [Background] Halder I, Shriver M, Thomas M, Fernandez JR, Frudakis T. A panel of ancestry informative markers for estimating individual biogeographical ancestry and admixture from four continents: utility and applications. Hum Mutat. 2008 May;29(5):648-58. doi: 10.1002/humu.20695. PMID 18286470
- [Background] Halloran BP, Bikle DD, Levens MJ, Castro ME, Globus RK, Holton E. Chronic 1,25-dihydroxyvitamin D3 administration in the rat reduces the serum concentration of 25-hydroxyvitamin D by increasing metabolic clearance rate. J Clin Invest. 1986 Sep;78(3):622-8. doi: 10.1172/JCI112619. PMID 3489007
- [Background] Harris SS, Dawson-Hughes B. Seasonal changes in plasma 25-hydroxyvitamin D concentrations of young American black and white women. Am J Clin Nutr. 1998 Jun;67(6):1232-6. doi: 10.1093/ajcn/67.6.1232. PMID 9625098
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Holick MF. Photobiology of Vitamin D. In: Pike JW, Glorieux FH, eds. Vitamin D. Vol 1. 2nd ed: Elsevier Academic Press; 2005:37-46.
- [Background] Hollis BW, Pittard WB 3rd. Evaluation of the total fetomaternal vitamin D relationships at term: evidence for racial differences. J Clin Endocrinol Metab. 1984 Oct;59(4):652-7. doi: 10.1210/jcem-59-4-652. PMID 6090493
- [Background] Horst RL. Exogenous versus endogenous recovery of 25-hydroxyvitamins D2 and D3 in human samples using high-performance liquid chromatography and the DiaSorin LIAISON Total-D Assay. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):180-2. doi: 10.1016/j.jsbmb.2010.03.010. Epub 2010 Mar 7. PMID 20214981
- [Background] Institute of Medicine (US) Committee to Review Dietary Reference Intakes for Vitamin D and Calcium; Ross AC, Taylor CL, Yaktine AL, Del Valle HB, editors. Dietary Reference Intakes for Calcium and Vitamin D. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK56070/ PMID 21796828
- [Background] Jacob AI, Sallman A, Santiz Z, Hollis BW. Defective photoproduction of cholecalciferol in normal and uremic humans. J Nutr. 1984 Jul;114(7):1313-9. doi: 10.1093/jn/114.7.1313. PMID 6330321
- [Background] Jin SE, Park JS, Kim CK. Pharmacokinetics of oral calcitriol in healthy human based on the analysis with an enzyme immunoassay. Pharmacol Res. 2009 Jul;60(1):57-60. doi: 10.1016/j.phrs.2009.03.005. Epub 2009 Mar 17. PMID 19427587
- [Background] Jurutka PW, Remus LS, Whitfield GK, Thompson PD, Hsieh JC, Zitzer H, Tavakkoli P, Galligan MA, Dang HT, Haussler CA, Haussler MR. The polymorphic N terminus in human vitamin D receptor isoforms influences transcriptional activity by modulating interaction with transcription factor IIB. Mol Endocrinol. 2000 Mar;14(3):401-20. doi: 10.1210/mend.14.3.0435. PMID 10707958
- [Background] Karohl C, Su S, Kumari M, Tangpricha V, Veledar E, Vaccarino V, Raggi P. Heritability and seasonal variability of vitamin D concentrations in male twins. Am J Clin Nutr. 2010 Dec;92(6):1393-8. doi: 10.3945/ajcn.2010.30176. Epub 2010 Oct 13. PMID 20943799
- [Background] Kleerekoper M, Nelson DA, Peterson EL, Flynn MJ, Pawluszka AS, Jacobsen G, Wilson P. Reference data for bone mass, calciotropic hormones, and biochemical markers of bone remodeling in older (55-75) postmenopausal white and black women. J Bone Miner Res. 1994 Aug;9(8):1267-76. doi: 10.1002/jbmr.5650090817. PMID 7976509
- [Background] Kleuser B, Cuvillier O, Spiegel S. 1Alpha,25-dihydroxyvitamin D3 inhibits programmed cell death in HL-60 cells by activation of sphingosine kinase. Cancer Res. 1998 May 1;58(9):1817-24. PMID 9581819
- [Background] Lips P, Duong T, Oleksik A, Black D, Cummings S, Cox D, Nickelsen T. A global study of vitamin D status and parathyroid function in postmenopausal women with osteoporosis: baseline data from the multiple outcomes of raloxifene evaluation clinical trial. J Clin Endocrinol Metab. 2001 Mar;86(3):1212-21. doi: 10.1210/jcem.86.3.7327. PMID 11238511
- [Background] Looker AC. Body fat and vitamin D status in black versus white women. J Clin Endocrinol Metab. 2005 Feb;90(2):635-40. doi: 10.1210/jc.2004-1765. Epub 2004 Nov 16. PMID 15546897
- [Background] Lore F, Di Cairano G, Periti P, Caniggia A. Effect of the administration of 1,25-dihydroxyvitamin D3 on serum levels of 25-hydroxyvitamin D in postmenopausal osteoporosis. Calcif Tissue Int. 1982;34(6):539-41. doi: 10.1007/BF02411300. PMID 6819073
- [Background] Lou YR, Molnar F, Perakyla M, Qiao S, Kalueff AV, St-Arnaud R, Carlberg C, Tuohimaa P. 25-Hydroxyvitamin D(3) is an agonistic vitamin D receptor ligand. J Steroid Biochem Mol Biol. 2010 Feb 15;118(3):162-70. doi: 10.1016/j.jsbmb.2009.11.011. Epub 2009 Nov 26. PMID 19944755
- [Background] Matsuoka LY, Wortsman J, Chen TC, Holick MF. Compensation for the interracial variance in the cutaneous synthesis of vitamin D. J Lab Clin Med. 1995 Nov;126(5):452-7. PMID 7595030
- [Background] Mawer EB, Schaefer K, Lumb GA, Stanbury SW. The metabolism of isotopically labelled vitamin D3 in man: the influence of the state of vitamin D nutrition. Clin Sci. 1971 Jan;40(1):39-53. doi: 10.1042/cs0400039. No abstract available. PMID 4321723
- [Background] Meyer MB, Goetsch PD, Pike JW. A downstream intergenic cluster of regulatory enhancers contributes to the induction of CYP24A1 expression by 1alpha,25-dihydroxyvitamin D3. J Biol Chem. 2010 May 14;285(20):15599-15610. doi: 10.1074/jbc.M110.119958. Epub 2010 Mar 17. PMID 20236932
- [Background] Miller B, Norman AW. Evidence for circadian rhythms in the serum levels of the vitamin D-dependent calcium-binding protein and in the activity of the 25-hydroxyvitamin D3-1-alpha-hydroxylase in the chick: studies on the mode of action of calciferol. FEBS Lett. 1982 May 17;141(2):242-4. doi: 10.1016/0014-5793(82)80057-4. No abstract available. PMID 7095152
- [Background] Nelson DA, Beck TJ, Wu G, Lewis CE, Bassford T, Cauley JA, LeBoff MS, Going SB, Chen Z. Ethnic differences in femur geometry in the women's health initiative observational study. Osteoporos Int. 2011 May;22(5):1377-88. doi: 10.1007/s00198-010-1349-4. Epub 2010 Aug 25. PMID 20737265
- [Background] Neuhouser ML, Wassertheil-Smoller S, Thomson C, Aragaki A, Anderson GL, Manson JE, Patterson RE, Rohan TE, van Horn L, Shikany JM, Thomas A, LaCroix A, Prentice RL. Multivitamin use and risk of cancer and cardiovascular disease in the Women's Health Initiative cohorts. Arch Intern Med. 2009 Feb 9;169(3):294-304. doi: 10.1001/archinternmed.2008.540. PMID 19204221
- [Background] Norman AW, Miller BE, Putkey JA. Evaluation of the diurnal production of 1,25-dihydroxyvitamin D and vitamin D's effects on intestinal membrane organization. Prog Biochem Pharmacol. 1980;17:160-7. No abstract available. PMID 6894193
- [Background] Raimondi S, Johansson H, Maisonneuve P, Gandini S. Review and meta-analysis on vitamin D receptor polymorphisms and cancer risk. Carcinogenesis. 2009 Jul;30(7):1170-80. doi: 10.1093/carcin/bgp103. Epub 2009 Apr 29. PMID 19403841
- [Background] Roff A, Wilson RT. A novel SNP in a vitamin D response element of the CYP24A1 promoter reduces protein binding, transactivation, and gene expression. J Steroid Biochem Mol Biol. 2008 Nov;112(1-3):47-54. doi: 10.1016/j.jsbmb.2008.08.009. Epub 2008 Sep 6. PMID 18824104
- [Background] Rohan TE, Negassa A, Chlebowski RT, Ceria-Ulep CD, Cochrane BB, Lane DS, Ginsberg M, Wassertheil-Smoller S, Page DL. A randomized controlled trial of calcium plus vitamin D supplementation and risk of benign proliferative breast disease. Breast Cancer Res Treat. 2009 Jul;116(2):339-50. doi: 10.1007/s10549-008-0213-0. Epub 2008 Oct 14. PMID 18853250
- [Background] Ross AC. The 2011 report on dietary reference intakes for calcium and vitamin D. Public Health Nutr. 2011 May;14(5):938-9. doi: 10.1017/S1368980011000565. No abstract available. PMID 21492489
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] Sathyapalan T, Shepherd J, Arnett C, Coady AM, Kilpatrick ES, Atkin SL. Atorvastatin increases 25-hydroxy vitamin D concentrations in patients with polycystic ovary syndrome. Clin Chem. 2010 Nov;56(11):1696-700. doi: 10.1373/clinchem.2010.144014. Epub 2010 Sep 3. PMID 20817794
- [Background] Stolzenberg-Solomon RZ, Hayes RB, Horst RL, Anderson KE, Hollis BW, Silverman DT. Serum vitamin D and risk of pancreatic cancer in the prostate, lung, colorectal, and ovarian screening trial. Cancer Res. 2009 Feb 15;69(4):1439-47. doi: 10.1158/0008-5472.CAN-08-2694. Epub 2009 Feb 10. PMID 19208842
- [Background] Stolzenberg-Solomon RZ, Vieth R, Azad A, Pietinen P, Taylor PR, Virtamo J, Albanes D. A prospective nested case-control study of vitamin D status and pancreatic cancer risk in male smokers. Cancer Res. 2006 Oct 15;66(20):10213-9. doi: 10.1158/0008-5472.CAN-06-1876. PMID 17047087
- [Background] Talwar SA, Aloia JF, Pollack S, Yeh JK. Dose response to vitamin D supplementation among postmenopausal African American women. Am J Clin Nutr. 2007 Dec;86(6):1657-62. doi: 10.1093/ajcn/86.5.1657. PMID 18065583
- [Background] Tang C, Chen N, Wu M, Yuan H, Du Y. Fok1 polymorphism of vitamin D receptor gene contributes to breast cancer susceptibility: a meta-analysis. Breast Cancer Res Treat. 2009 Sep;117(2):391-9. doi: 10.1007/s10549-008-0262-4. Epub 2009 Jan 6. PMID 19145484
- [Background] Tarcin O, Yavuz DG, Ozben B, Telli A, Ogunc AV, Yuksel M, Toprak A, Yazici D, Sancak S, Deyneli O, Akalin S. Effect of vitamin D deficiency and replacement on endothelial function in asymptomatic subjects. J Clin Endocrinol Metab. 2009 Oct;94(10):4023-30. doi: 10.1210/jc.2008-1212. Epub 2009 Jul 7. PMID 19584181
- [Background] Thieden E, Jorgensen HL, Jorgensen NR, Philipsen PA, Wulf HC. Sunbed radiation provokes cutaneous vitamin D synthesis in humans--a randomized controlled trial. Photochem Photobiol. 2008 Nov-Dec;84(6):1487-92. doi: 10.1111/j.1751-1097.2008.00372.x. Epub 2008 May 29. PMID 18513233
- [Background] Trivedi DP, Doll R, Khaw KT. Effect of four monthly oral vitamin D3 (cholecalciferol) supplementation on fractures and mortality in men and women living in the community: randomised double blind controlled trial. BMJ. 2003 Mar 1;326(7387):469. doi: 10.1136/bmj.326.7387.469. PMID 12609940
- [Background] Uitterlinden AG, Fang Y, Van Meurs JB, Pols HA, Van Leeuwen JP. Genetics and biology of vitamin D receptor polymorphisms. Gene. 2004 Sep 1;338(2):143-56. doi: 10.1016/j.gene.2004.05.014. PMID 15315818
- [Background] Wactawski-Wende J, Kotchen JM, Anderson GL, Assaf AR, Brunner RL, O'Sullivan MJ, Margolis KL, Ockene JK, Phillips L, Pottern L, Prentice RL, Robbins J, Rohan TE, Sarto GE, Sharma S, Stefanick ML, Van Horn L, Wallace RB, Whitlock E, Bassford T, Beresford SA, Black HR, Bonds DE, Brzyski RG, Caan B, Chlebowski RT, Cochrane B, Garland C, Gass M, Hays J, Heiss G, Hendrix SL, Howard BV, Hsia J, Hubbell FA, Jackson RD, Johnson KC, Judd H, Kooperberg CL, Kuller LH, LaCroix AZ, Lane DS, Langer RD, Lasser NL, Lewis CE, Limacher MC, Manson JE; Women's Health Initiative Investigators. Calcium plus vitamin D supplementation and the risk of colorectal cancer. N Engl J Med. 2006 Feb 16;354(7):684-96. doi: 10.1056/NEJMoa055222. PMID 16481636
- [Background] Williams GM, Hard GC. Correspondence re: R. R. Love, The National Surgical Adjuvant Breast Project (NSABP) Breast Cancer Prevention Trial revisited. Cancer Epidemiol., Biomarkers & Prev., 2: 403-407, 1993. Cancer Epidemiol Biomarkers Prev. 1994 Mar;3(2):185-6. No abstract available. PMID 8049643
- [Background] Wilson RT, Chase GA, Chrischilles EA, Wallace RB. Hip fracture risk among community-dwelling elderly people in the United States: a prospective study of physical, cognitive, and socioeconomic indicators. Am J Public Health. 2006 Jul;96(7):1210-8. doi: 10.2105/AJPH.2005.077479. Epub 2006 May 30. PMID 16735617
- [Background] Wilson RT, Roff AN, Dai PJ, Fortugno T, Douds J, Chen G, Grove GL, Nikiforova SO, Barnholtz-Sloan J, Frudakis T, Chinchilli VM, Hartman TJ, Demers LM, Shriver MD, Canfield VA, Cheng KC. Genetic Ancestry, Skin Reflectance and Pigmentation Genotypes in Association with Serum Vitamin D Metabolite Balance. Horm Mol Biol Clin Investig. 2011 Sep;7(1):279-293. doi: 10.1515/HMBCI.2011.021. PMID 23525585
- [Background] Xu HM, Tepper CG, Jones JB, Fernandez CE, Studzinski GP. 1,25-Dihydroxyvitamin D3 protects HL60 cells against apoptosis but down-regulates the expression of the bcl-2 gene. Exp Cell Res. 1993 Dec;209(2):367-74. doi: 10.1006/excr.1993.1322. PMID 8262155